CLINICAL TRIAL: NCT02329743
Title: A Multicenter, Double-Masked, Parallel-Group, Vehicle-Controlled Study to Assess the Efficacy and Safety of RX-10045 Nanomicellar Ophthalmic Solution for Treatment of Ocular Inflammation and Pain in Subjects Undergoing Cataract Surgery
Brief Title: Efficacy and Safety of RX-10045 Ophthalmic Solution for Ocular Inflammation and Pain in Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: A.T. Resolve SARL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATR-45-1401
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Inflammation; Pain; Cataract
MeSH Terms: conditions — Inflammation; Pain; Cataract | interventions — isopropyl 5,12-hydroxypentadeca-8,10-dien-6,14-diynoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- RX-10045 0.05% nanomicellar solution (Experimental): topical eye drops
  Interventions: Drug: RX-10045
- RX-10045 0.1% nanomicellar solution (Experimental): topical eye drops
  Interventions: Drug: RX-10045
- Vehicle (Placebo Comparator): topical eye drops
  Interventions: Drug: RX-10045

INTERVENTIONS:
Drug: RX-10045 — topical therapy

SUMMARY:
The primary objective of this study is to assess the efficacy and safety of 2 concentrations of RX-10045 ophthalmic solution, 0.05% and 0.1%, compared to placebo for the treatment of ocular inflammation and pain in subjects undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cataract surgery (phacoemulsification or extracapsular extraction) with posterior chamber intraocular lens implantation in the capsular bag.

Exclusion Criteria:

* Any additional surgical procedures at the time of the cataract surgery
* Refractive surgery in the study eye within the past 2 years
* History or presence of noninfectious inflammatory ocular disease (e.g., episcleritis, scleritis, uveitis) in either eye
* Intraocular pressure of > 21 mm Hg in either eye
* Proliferative or severe nonproliferative diabetic retinopathy in either eye
* Neovascular/wet age-related macular degeneration in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Sablinski, MD, Study Director — Auven Therapeutics
Locations (1):
- Auven Therapeutics, Murray Hill, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RX-10045 0.05% Nanomicellar Solution | RX-10045 0.1% Nanomicellar Solution | Vehicle
Started | 84 | 87 | 85
Completed | 78 | 80 | 77
Not Completed | 6 | 7 | 8
Not completed — Adverse Event | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4 | 1
Not completed — Other | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RX-10045 0.05% Nanomicellar Solution | RX-10045 0.1% Nanomicellar Solution | Vehicle | Total
Number analyzed (Participants) | 79 | 79 | 78 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.2) | 66.2 (8.6) | 66.1 (8.9) | 66.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 48 | 138
  Male | 37 | 31 | 30 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 7 | 30
  Not Hispanic or Latino | 67 | 68 | 71 | 206
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 2 | 1 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 4 | 5
  Black or African American | 7 | 7 | 6 | 20
  White | 67 | 67 | 63 | 197
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Clearing of Anterior Inflammation
Description: score of zero for the Standardization of Uveitis Nomenclature scale
Time Frame: Day 8
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | RX-10045 0.05% Nanomicellar Solution | RX-10045 0.1% Nanomicellar Solution | Vehicle
Number analyzed (Participants) | 79 | 79 | 78
Participants | 18 | 18 | 13

2. Secondary Outcome: Proportion of Subjects Reporting no Ocular Pain
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | RX-10045 0.05% Nanomicellar Solution | RX-10045 0.1% Nanomicellar Solution | Vehicle
Number analyzed (Participants) | 79 | 79 | 78
Participants | 25 | 21 | 33

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | RX-10045 0.05% Nanomicellar Solution | RX-10045 0.1% Nanomicellar Solution | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/79 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/78
Other Adverse Events (participants affected / at risk) | 0/79 | 0/79 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No